CLINICAL TRIAL: NCT05383898
Title: A Phase 1/2, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of D-1553 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Study to Evaluate D-1553 in Subjects With Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D1553-102
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a Dose escalation of D-1553 (Experimental): Phase 1a will evaluate up to sequential cohorts with different doses of D-1553 to determine safety, tolerability, MTD and RDE in patients with solid tumors with KRasG12C mutation
  Interventions: Drug: D-1553
- Phase 1b Dose expansion of D-1553 (Experimental): Phase 1b will evaluate more subjects with up to 2 different doses of D-1553 to confirm the recommended phase 2 dose.
  Interventions: Drug: D-1553
- Phase 2 of D-1553 monotherapy (Experimental): Phase 1b will evaluate more subjects at the recommended phase 2 dose of D-1553 to evaluate the efficacy.
  Interventions: Drug: D-1553

INTERVENTIONS:
Drug: D-1553 — D-1553 is a novel, targeted KRasG12C inhibitor that is being developed as a potential oral agent for advanced or metastatic solid tumors with KRasG12C mutation.

SUMMARY:
This is a phase 1/2, open label study of D-1553 single agent treatment to assess the safety and tolerability, identify the MTD and RP2D, evaluate the PK properties and antitumor activities in subjects with advanced or metastatic NSCLC with KRasG12C mutation

ELIGIBILITY:
Inclusion Criteria:

* Subject with histologically proven, locally advanced, unresectable and/or metastatic NSCLC for which no standard treatment is available or the subject is refractory to or intolerant of existing standard treatment.
* Subject has KRasG12C mutation in tumor tissue or other biospecimens containing cancer cells or DNA. Historical, local laboratory result (up to 5 years prior to this study) can be used for Phase 1 subjects. Phase 2 subjects must be tested for KRasG12C mutation by a central laboratory.
* Subject has measurable disease according to RECIST, v1.1

Exclusion Criteria:

* Subject with unstable or progressive central nervous system (CNS) metastases.
* Subjects with clinically significant cardiovascular disease
* Subject with interstitial lung disease (ILD) or any active systemic infection including but not limited to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Subject has impaired gastrointestinal (GI) function or GI diseases that may significantly alter the absorption or metabolism of oral medications.
* Subject is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Subject incidence of Dose-limiting toxicities (DLT) | through out the DLT period, approximately 21 days
  Subject incidence of Dose-limiting toxicities (DLT)
Number of subjects participants with adverse events | Through study completion, approximately 3 years
  Number of subjects participants with adverse events
antitumor activity of D-1553 in subjects with advanced or metastatic NSCLC with KRASG12C mutation | Through study completion, approximately 3 years
  Overall Response Rate (ORR, Complete Response [CR] + Partial Response [PR])

SECONDARY OUTCOMES:
Plasma concentration of D-1553 | approximately 6 months
  Plasma concentration of D-1553 as a single agent in subjects with advanced or metastatic NSCLC with KRas G12C mutation

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (2):
- China (2):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Cancer Hospital of the University of Chinese Academy of Sciences,, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song Z, Li Z, Zhang Y, Wang P, Jiang L, Zhao Y, Zhou J, Wang X, Zhuang W, Shi J, Huang D, Dang X, Cang S, Gong Y, Jin S, Li W, Dong X, Zhang J, Zhao M, Meng X, Liu X, Fang J, Wu P, Lu J, Zhang L, Yang J, Wang X, Luo H, Cui J, Zhang Z, Wang J, Li G, Wu L, Yu Y, Fang Y, Lv D, Yang W, Chen L, Yang N, Li K, Ma R, Wang M, Zhou H, Hu S, Li Q, Zhuang Z, Cao B, Zhu W, Xu C, Wang W, Xiang Z, Shi Z, Wang Y, Zhang L, Lu S. Garsorasib in patients with KRAS G12C-mutated non-small-cell lung cancer: A pooled analysis of phase 1/2 study. Eur J Cancer. 2026 Jan;232:116153. doi: 10.1016/j.ejca.2025.116153. Epub 2025 Nov 29. PMID 41330054
- [Derived] Li Z, Dang X, Huang D, Jin S, Li W, Shi J, Wang X, Zhang Y, Song Z, Zhang J, Zhuang W, Liu X, Jiang L, Meng X, Zhao M, Zhou J, Zhang L, Wang P, Luo H, Yang J, Cang S, Wang X, Zhang L, Lu S; D1553-102 Study Group. Garsorasib in patients with KRASG12C-mutated non-small-cell lung cancer in China: an open-label, multicentre, single-arm, phase 2 trial. Lancet Respir Med. 2024 Aug;12(8):589-598. doi: 10.1016/S2213-2600(24)00110-3. Epub 2024 Jun 10. PMID 38870979
- [Derived] Li Z, Song Z, Zhao Y, Wang P, Jiang L, Gong Y, Zhou J, Jian H, Dong X, Zhuang W, Cang S, Yang N, Fang J, Shi J, Lu J, Ma R, Wu P, Zhang Y, Song M, Xu CW, Shi Z, Zhang L, Wang Y, Wang X, Zhang Y, Lu S. D-1553 (Garsorasib), a Potent and Selective Inhibitor of KRASG12C in Patients With NSCLC: Phase 1 Study Results. J Thorac Oncol. 2023 Jul;18(7):940-951. doi: 10.1016/j.jtho.2023.03.015. Epub 2023 Mar 21. PMID 36948246